CLINICAL TRIAL: NCT07030985
Title: Perfusion Imaging Score to Predict Delayed Cerebral Ischemia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Anna Maria Bombardieri, Clinical Associate Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 81412
Record Dates: First submitted 2025-06-12; First posted 2025-06-22 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Aneurysmal Subarachnoid Hemorrhage; Cerebral Ischemia
Keywords: computed tomography perfusion; brain perfusion; early detection; prediction
MeSH Terms: conditions — Subarachnoid Hemorrhage; Brain Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients diagnosed with aSAH (Experimental): Patients will undergo the following study procedures:
  * a CTP scan after aSAH diagnosis
  * neurological and the neuropsychological tests at 12-month after the hemorrhage.
  Interventions: Radiation: CTP scan; Diagnostic Test: Neurological and neuropsychological testing

INTERVENTIONS:
Radiation: CTP scan — Patients with diagnosed aSAH and no evidence of early radiologic vasospasm will receive a CTP scan within 48 hours of aSAH symptom onset.
Diagnostic Test: Neurological and neuropsychological testing — All enrolled patients will receive neurological and neuropsychological assessment at 12 months after aSAH.

SUMMARY:
Aneurysmal subarachnoid hemorrhage (aSAH) is a significant public health concern, annually affecting over 30,000 Americans and ranking among the leading causes of stroke-related life-years lost in individuals aged 65 and younger. Delayed cerebral ischemia (DCI), occurring in 20% to 40% of aSAH survivors, is a major contributor to brain injury and disability. Timely recognition of DCI is crucial for improving neurological outcomes and preventing irreversible cerebral infarction. However, current methods have substantial limitations, hindering early and reliable detection. This proposal seeks to address these challenges through determining the ability of perfusion imaging to predict DCI and correlate with neurological and neuropsychological outcomes.

DETAILED DESCRIPTION:
Patients with a diagnosis of aSAH and no early radiologic vasospasm on admission demonstrated by DSA will receive a CT Perfusion (CTP) scan within 48 hours of aSAH symptom onset. The researchers seek to determine whether these baseline scans will identify perfusion parameters predictive of DCI. At 12-months mark post-hemorrhage, neurological and neuropsychological tests will be conducted to determine whether perfusion imaging correlates with neurological and neuropsychological outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years with a diagnosis of aSAH

Exclusion Criteria:

* chronic kidney disease stage IV
* pregnancy
* allergy to iodine that precludes CTP
* subjects with significant aphasia, blindness, or other factors that limit their participation in the cognitive assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Delayed Cerebral Ischemia (DCI) | During hospitalization (within 14 days of aneurysmal subarachnoid hemorrhage (aSAH))
  DCI will be diagnosed using the 2010 consensus definition, including new focal neurological impairments (e.g., hemiparesis, aphasia, apraxia, hemianopia, or neglect) or a decrease of ≥2 points on the Glasgow Coma Scale lasting ≥1 hour, not immediately after aneurysm treatment and not due to other identifiable causes.

SECONDARY OUTCOMES:
Correlation Between Baseline Perfusion Parameters and 12-Month Neurological Outcome | 12 months post-aSAH
  Assessment of whether poor baseline perfusion profile (DCI Index Score (DIS) > 0.06) correlates with worse outcomes on neurological and neuropsychological assessments including modified Rankin Scale (mRS), 36-Item Short Form Health Survey (SF-36), and standardized cognitive test z-scores.
Modified Rankin Scale (mRS) | 12 months post-aSAH
  Measurement of functional disability using mRS, categorized as favorable (0-3) or unfavorable (4-6), to assess long-term disability and its association with baseline perfusion.
Health-Related Quality of Life (HRQoL, SF-36) | 12 months post-aSAH
  HRQoL will be reported as standardized z-scores, with higher scores indicating better performance.
Global Mental Status - Montreal Cognitive Assessment (MoCA) | 12 months post-aSAH
  Screens for mild cognitive impairment across multiple cognitive domains. Raw scores range from 0 to 30. Favorable outcome: MoCA score ≥ 26, unfavorable outcome: MoCA score < 26 (suggestive of cognitive impairment).
Executive Functioning - Wisconsin Card Sorting Test (WCST) | 12 months post-aSAH
  Measures executive functioning, including cognitive flexibility and problem-solving. The number of categories completed and total errors will be converted to age-adjusted z-scores.
  Favorable outcome: z-score ≥ -1.0, unfavorable outcome: z-score < -1.0 (indicative of cognitive impairment in executive functioning).
Processing Speed - Symbol Digit Modalities Test (SDMT) | 12 months post-aSAH
  Assesses visual scanning, tracking, and motor speed. Raw scores are adjusted for age and converted to z-scores. Favorable outcome: z-score ≥ -1.0, unfavorable outcome: z-score < -1.0
Language - Boston Naming Test (BNT) | 12 months post-aSAH
  Evaluates confrontational word retrieval and naming ability. Scores are standardized using age norms. Favorable outcome: z-score ≥ -1.0, unfavorable outcome: z-score < -1.0
Verbal Fluency - FAS Test | 12 months post-aSAH
  Tests lexical fluency by asking participants to generate words beginning with F, A, and S in a set time period. Z-scores are calculated from age-adjusted norms. Favorable outcome: z-score ≥ -1.0, unfavorable outcome: z-score < -1.0
Memory - Hopkins Verbal Learning Test-Revised (HVLT-R) | 12 months post-aSAH
  Assesses verbal learning and memory, including immediate recall, delayed recall, and recognition. Performance is normed and converted into z-scores. Favorable outcome: z-score ≥ -1.0, unfavorable outcome: z-score < -1.0
Composite Neuropsychological Test Scores | 12 months post-aSAH
  Analysis of cognitive function via composite z-scores derived from tests across executive function, memory, language, verbal fluency, processing speed, and global cognition (e.g., MoCA, HVLT-R, Boston Naming Test). Worse outcomes are defined by lower neuropsychological z-scores.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dodd WS, Laurent D, Dumont AS, Hasan DM, Jabbour PM, Starke RM, Hosaka K, Polifka AJ, Hoh BL, Chalouhi N. Pathophysiology of Delayed Cerebral Ischemia After Subarachnoid Hemorrhage: A Review. J Am Heart Assoc. 2021 Aug 3;10(15):e021845. doi: 10.1161/JAHA.121.021845. Epub 2021 Jul 30. PMID 34325514
- [Background] Macdonald RL. Delayed neurological deterioration after subarachnoid haemorrhage. Nat Rev Neurol. 2014 Jan;10(1):44-58. doi: 10.1038/nrneurol.2013.246. Epub 2013 Dec 10. PMID 24323051
- [Background] Rowland MJ, Hadjipavlou G, Kelly M, Westbrook J, Pattinson KT. Delayed cerebral ischaemia after subarachnoid haemorrhage: looking beyond vasospasm. Br J Anaesth. 2012 Sep;109(3):315-29. doi: 10.1093/bja/aes264. PMID 22879655
- [Background] Baumgartner RW. Transcranial color duplex sonography in cerebrovascular disease: a systematic review. Cerebrovasc Dis. 2003;16(1):4-13. doi: 10.1159/000070108. PMID 12766355
- [Background] Nguyen AM, Williamson CA, Pandey AS, Sheehan KM, Rajajee V. Screening Computed Tomography Angiography to Identify Patients at Low Risk for Delayed Cerebral Ischemia Following Aneurysmal Subarachnoid Hemorrhage. Front Neurol. 2021 Nov 12;12:740241. doi: 10.3389/fneur.2021.740241. eCollection 2021. PMID 34867722
- [Background] Mir DI, Gupta A, Dunning A, Puchi L, Robinson CL, Epstein HA, Sanelli PC. CT perfusion for detection of delayed cerebral ischemia in aneurysmal subarachnoid hemorrhage: a systematic review and meta-analysis. AJNR Am J Neuroradiol. 2014 May;35(5):866-71. doi: 10.3174/ajnr.A3787. Epub 2013 Dec 5. PMID 24309123
- [Background] Starnoni D, Maduri R, Hajdu SD, Pierzchala K, Giammattei L, Rocca A, Grosfilley SB, Saliou G, Messerer M, Daniel RT. Early Perfusion Computed Tomography Scan for Prediction of Vasospasm and Delayed Cerebral Ischemia After Aneurysmal Subarachnoid Hemorrhage. World Neurosurg. 2019 Oct;130:e743-e752. doi: 10.1016/j.wneu.2019.06.213. Epub 2019 Jul 5. PMID 31284055
- [Background] Bashir A, Andresen M, Bartek J Jr, Cortsen M, Eskesen V, Wagner A. Intra-arterial nimodipine for cerebral vasospasm after subarachnoid haemorrhage: Influence on clinical course and predictors of clinical outcome. Neuroradiol J. 2016 Feb;29(1):72-81. doi: 10.1177/1971400915626429. Epub 2016 Jan 29. PMID 26825134
- [Background] Dorhout Mees SM, Rinkel GJ, Feigin VL, Algra A, van den Bergh WM, Vermeulen M, van Gijn J. Calcium antagonists for aneurysmal subarachnoid haemorrhage. Cochrane Database Syst Rev. 2007 Jul 18;2007(3):CD000277. doi: 10.1002/14651858.CD000277.pub3. PMID 17636626
- [Background] Hosmann A, Rauscher S, Wang WT, Dodier P, Bavinzski G, Knosp E, Gruber A. Intra-Arterial Papaverine-Hydrochloride and Transluminal Balloon Angioplasty for Neurointerventional Management of Delayed-Onset Post-Aneurysmal Subarachnoid Hemorrhage Vasospasm. World Neurosurg. 2018 Nov;119:e301-e312. doi: 10.1016/j.wneu.2018.07.138. Epub 2018 Jul 24. PMID 30053563